CLINICAL TRIAL: NCT04145518
Title: Mechanistic Characterization of Uterine Pain (MCUP) to Improve Diagnosis and Treatment for Dysmenorrhea
Brief Title: Mechanistic Characterization of Uterine Pain
Acronym: MCUP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kevin Hellman, Research Associate Professor, Endeavor Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: EH19-040; R01HD098193-01A1 (NIH)
Record Dates: First submitted 2019-10-25; First posted 2019-10-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Dysmenorrhea (Disorder); Dysmenorrhea Primary; Dysmenorrhea Secondary; Endometrial Diseases; Leiomyoma; Fibroid Uterus
Keywords: pain; NSAID; women's health; uterus; MRI
MeSH Terms: conditions — Dysmenorrhea; Uterine Diseases; Leiomyoma; Pain | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Naproxen/Placebo Crossover (Active Comparator): Participants will be randomized to take either a placebo pill or a single 550 mg naproxen sodium pill. Randomization with a block size only known by the statistician, will be programmed to be allocated out of REDcap.
  Our clinical research pharmacy will provide naproxen and an identical looking placebo in containers with codes only known to the statistician to provide a double-blinded experimental design.
  On a subsequent episode of menstrual pain (1-2 months later), participants will receive the opposite treatment and undergo the exact same assessments.
  Interventions: Drug: Naproxen Sodium
- Placebo/Naproxen Crossover (Placebo Comparator): Participants will receive placebo first in this arm.
  Interventions: Drug: Naproxen Sodium

INTERVENTIONS:
Drug: Naproxen Sodium — Participants will be randomized to take either a placebo pill or a single 550 mg naproxen sodium pill.
  Other Names: Placebo

SUMMARY:
There are limited treatment options for management of dysmenorrhea, and the physiological processes they affect are not completely understood. For example, NSAIDs are effective in reducing menstrual pain in some women by inhibition of prostaglandin synthesis, but whether those effects are mediated by affecting contractility, perfusion, or hypoxemia is unknown. Understanding how these drugs relieve menstrual pain (and why they fail) would be of substantial clinical significance. Given the foregoing, Two Specific Aims are proposed:

Aim #1: Characterize menstrual pain phenotypes associated with impairments in myometrial activity, perfusion, and/or oxygenation. Continuous MRI scans of the uterus will be performed with simultaneous measurement of self-reported pain in healthy women and those experiencing menstrual pain. The investigators will include cohorts of women with imaging diagnosed leiomyoma and surgically-confirmed endometriosis to evaluate the contribution of structurally identifiable factors. Based on preliminary data, the investigators anticipate finding four phenotypes with menstrual pain related to: 1) myometrial activity, 2) inadequate perfusion and/or oxygenation, 3) a combination of phenotypes 1 & 2, and 4) a non-uterine source.

Aim #2: Evaluate the effects of naproxen on myometrial activity, perfusion, and/or oxygenation with respect to pain relief. In women with primary dysmenorrhea, the investigators will acquire pelvic MRI scans and evaluate self-reported menstrual cramping pain before and after administration of randomized naproxen or placebo.

Naproxen could principally affect one or more potential sources of uterine pain such as myometrial activity, perfusion, and/or oxygenation. The investigators will corroborate preliminary data findings, which suggest menstrual phenotypes with myometrial activity will be more likely to respond. Conversely, Aim 2 will also elucidate the mechanisms responsible for inadequate pain relief from naproxen.

Bioavailability of naproxen levels and other molecules associated with NSAID-resistance will be evaluated from the serum of participants after taking naproxen using HPLC-MS.

DETAILED DESCRIPTION:
Due to a lack of noninvasive tools to study uterine physiology, the root causes of menstrual cramping pain within primary dysmenorrhea and secondary dysmenorrhea (leiomyoma, endometriosis, adenomyosis) remain unknown. This pain does not respond to typical over-the-counter anti-inflammatories in 15% of women and is a leading risk factor for developing challenging chronic pelvic pain disorders. In order to guide drug discoveries and create personalized treatment approaches, it is essential to unveil the underlying mechanisms of dysmenorrhea. Our research program has focused on key gaps in our knowledge of uterine physiology, such as the contributions of uterine contractions, perfusion, and oxygenation to menstrual pain. Although these factors are strongly implicated in this debilitating pain disorder, confirmatory human data is still needed. Such research would be quite timely, as numerous drug candidates targeting these potential mechanisms already exist. Our collaborative team has developed MRI-based tools to noninvasively and dynamically measure uterine contractions, perfusion, relative tissue oxygenation, and metabolites indicative of anaerobic respiration. The investigators have also pioneered methods that link spontaneous pain report to simultaneous uterine events. Together, these methods will allow us to evaluate the contribution of contractility, perfusion, or hypoxemia to menstrual pain. Notably, our preliminary data supports our central hypothesis that menstrual pain is associated with different phenotypes involving myometrial hypercontractility, impaired uterine perfusion, uterine hypoxemia, or a non-uterine source. Since understanding how current anti-inflammatory medications relieve or prevent pain (and why they fail) is valuable for the development of improved treatment strategies, the investigators will also investigate the effects of naproxen on uterine physiology in women with menstrual pain. To test our hypothesized contributions of altered uterine muscle activity, perfusion, and oxygenation on pain, The investigators propose: Aim 1: Characterize menstrual pain phenotypes associated with impairments in myometrial activity, perfusion, and/or oxygenation. Continuous MRI sequences of the uterus will be performed with simultaneous measurement of self-reported pain in healthy women and those experiencing menstrual pain. A cohort of women with leiomyoma and endometriosis will also be analyzed to evaluate the contribution of myometrial activity, perfusion, and oxygenation in women with structurally identifiable conditions. Aim 2: Evaluate the effects of naproxen on myometrial activity, perfusion, and/or oxygenation with respect to pain relief. Preliminary data suggests unresolved myometrial activity and inadequate naproxen absorption are associated with insufficient pain relief. Evaluating the naproxen-dependent effects of uterine physiology will provide a foundation for diagnostic tests to indicate relevant personalized treatment for patients that have failed conventional treatments. Further translation of these studies could advance mechanisms for discovery in other chronic pelvic pain conditions and uterine disorders such as idiopathic preterm labor and unexplained infertility.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Primary Dysmenorrhea Group: All cases (n=70) will have pain in the region between the umbilicus and the perineum, above the level of the inguinal ligament, and rate their average pain greater than or equal to 6/10 (0 = no pain; 10 = worst imaginable pain) during menses when not using NSAIDs. The investigators will use strict inclusion criteria and verification with structural MRI to ensure patients with primary dysmenorrhea most likely do not have endometriosis, leiomyoma, or adenomyosis as described below. It is not possible to reliably evaluate superficial endometriosis with MRI (Nisenblat et al., 2016), but suspicious cases for deep infiltrating endometriosis will be confirmed by the radiologists who routinely evaluate MRIs for our gynecological surgical service. Although it is impossible to rule out endometriosis without surgery, in select cases The investigators will use clinical exams and criteria supported by decision trees (Eskenazi et al., 2001; Chapron et al., 2005, 2011; Vercellini et al., 2007) that suggest the detection of endometriosis stage 2 or higher would be unlikely (<15%) in this population. Participants with dysmenorrhea that rate their bowel pain, dyspareunia, or non-menstrual pelvic pain equal to or greater than 40 on 0-100 visual analog pain scale on the McGill Pain Questionnaire will be given the option to participate in an additional clinical exam visit. To reduce the likelihood of comorbid endometriosis, primary dysmenorrhea participants with symptoms of endometriosis described above, will be required to have a negative clinical exam and no immediate family history of endometriosis to qualify for final analyses.

Inclusion Criteria for Leiomyomata Group: The investigators will also study participants with leiomyomata (n=20) because it is a frequent cause of menstrual pain and will often be identified in disqualified primary dysmenorrhea participants. Leiomyomata (nondegenerated) will be diagnosed by foci homogeneously hypointense on T2, but isointense relative to myometrium on T1 according to standard definitions (Kubik-Huch et al., 2018). To reduce variability within this category, the investigators will restrict enrollment to small to medium sized intramural leiomyomata (30 to 150 cm3 combined volume). The investigators anticipate 10 participants with leiomyomata will be identified from incidental MRI during this study, while 10 more will be recruited from advertisements and our clinic. A smaller cohort is studied here because the main purpose of this group is to establish whether the physiological basis for menstrual pain in women with leiomyomata is significantly different than women with primary dysmenorrhea. Participants with leiomyomata, who are also symptomatic with surgically diagnosed endometriosis will be excluded.

Inclusion Criteria for Endometriosis Group: Participants without leiomyomata, but symptomatic for endometriosis (n=20) will be enrolled before planned surgical excision (follow-up surgery from an earlier diagnosis). The investigators will confirm a diagnosis of Stage 2, 3, or 4 endometriosis following surgery. For the patients without confirmed abnormal surgical findings for endometriosis with dysmenorrhea will be considered as primary dysmenorrhea cases. Dr. Tu's pelvic pain division performs over 100 laparoscopic pain evaluations annually (many with deep infiltrating disease) enabling us to characterize MRI signals in surgically confirmed endometriosis patients. A smaller cohort is studied here because the main purpose of this group is to establish whether the physiological basis for menstrual pain in women with endometriosis is significantly different than women with primary dysmenorrhea.

Inclusion Criteria for Healthy Controls: Healthy control cases (n=20) must rate their average menstrual pain < =2/10 over that past 6 months (without NSAID use) and have no other concurrent pain diagnoses or leiomyomata. Their lack of concurrent pain diagnoses will be confirmed with questionnaires (NIH PROMIS scales, Rome Foundation IBS criteria (Palsson et al., 2016), AUA bladder pain syndrome criteria (Hanno et. al. 2012), and the Complex Medical Symptom Inventory (Williams and Schilling, 2009) and a medical exam screen. Healthy controls and participants with primary dysmenorrhea will be ratio-metrically age-matched with comparable pregnancy history to ensure similar demographics between groups.

Exclusion Criteria:

Age restrictions for all study participants: Regularly menstruating women (age 18-45) will be identified using our well-tested community-wide recruitment strategy, including approaching our division's busy gynecological disorders clinic, and the departments of Ob/Gyn at NorthShore and the University of Chicago. Although women above the age of 45 can have menstrual pain, irregularities in perimenopause could cause confounding effects on uterine physiology and scheduling difficulty. Similarly, irregularities in menstruation, ovulation, and pain levels in participants under age 18 could potentially detract from meaningful interpretation of phenotypes (Seidman et al., 2018). Additionally, before age 18, the uterus is still developing and substantially increasing in size (Porcu et al., 1989; Verguts et al., 2013). Thus, to limit potential confounding effects, participants under the age of 18 will be investigated in a separate study.

Menstruation-related exclusion criteria for all study participants: The investigators will exclude certain participants with conditions associated with the absence of regular menses such as polycystic ovarian syndrome, pregnancy, current use of any continuous hormonal medication or contraceptive, or Asherman's syndrome.

MRI-related or participation related exclusion criteria for all study participants:

The investigators will exclude participants with criteria that would affect our ability to obtaining meaningful MRI data such as

1. presence of an intrauterine device (IUD). The use of an IUD potentially affects interpretability of MRI because it creates an imaging artifact in the endometrium extending to the myometrium.
2. inability to read or comprehend the informed consent written in English,
3. history of metallic implants,
4. history of metallic injury,
5. any diagnosed condition that would preclude investigation with MRI (e.g., claustrophobia),
6. BMI >40,
7. allergy or inability to tolerate naproxen

Exclusion criteria for known factors that affect the interpretability of the data for all study participants:

1. thyroid dysfunction,
2. adrenal dysfunction,
3. renal disorders,
4. liver disorders,
5. coagulopathy,
6. prolactinoma,
7. von Willebrand disease,
8. platelet disorders,
9. diabetic neuropathy,
10. gastrointestinal conditions or surgeries that would affect naproxen absorption,
11. active genitourinary or sexually transmitted infection

Provisional exclusion for primary analyses for all study participants: Acute or chronic conditions associated with pelvic pain with a defined anatomical cause other than endometriosis or leiomyoma (e.g., pathological ovarian cysts, significant persistent hydro/hematosalpinx, untreated pelvic inflammatory disease, active pelvic or abdominal malignancies, Mullerian anomalies, or stage 3 uterine prolapse), and comorbid diagnosis of significant leiomyoma and endometriosis.

Note: these exclusion criteria may be incidentally discovered after the MRI scan and confirmed with a radiologist's or Dr. Tu's diagnosis.

Provisional exclusion for adenomyosis group: Because the frequency of adenomyosis is low or unknown, and may consist of multiple subtypes resulting in heterogeneity and inadequate statistical power, adenomyosis patients are not a planned study group and diagnosed cases will be initially excluded from recruitment. Focal and diffuse adenomyosis will be excluded by guidelines (Chapron et al., 2017) adapted from the Kishi criteria (Kishi et al., 2012): maximal junctional zone thickness exceeding 12 mm, a ratio of junctional zone thickness to myometrium exceeding 40%, or high-intensity foci within the myometrium. If a substantial number of adenomyosis participants participate, as discovered after-the-fact with MRI, results will be analyzed.

Intermediate levels of dysmenorrhea pain exclusion: Participants with mild menstrual pain (between 3 and 5 on a 0-10 scale) will be excluded. Our prior experience with this cohort (Westling et al., 2013) suggests that The investigators may encounter a floor effect when studying the effectiveness of NSAIDs. Also, since this cohort is most likely to respond to NSAIDs, it is imperative The investigators study the mechanisms of the most severe sufferers of refractory menstrual pain.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must have a uterus and must not be undergoing hormone therapy.
Enrollment: 183 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Calculate response profiles of MRI signals for each menstrual pain phenotype | Initial Scan (1 hour)
  The investigators will calculate the change in R2*, ASL (arterial spin label), HASTE, and BOLD (Blood Oxygen Level Dependent) signal for each menstrual pain phenotype.
  Principal component analysis of derived MRI signal variables and subsequent scree plotting will be used to reduce the dataset to 4-6 representative parameters that meaningfully separate potential phenotypes via hierarchical cluster analysis (R cluster library). Cluster dissimilarity metrics will be used to establish the probable number of phenotypes. Thus, our analyses are not entirely dependent on hypothesized phenotypes. A post-hoc ANOVA will be performed on relevant signal intensity variables to validate differences between the phenotypes. A post-hoc ANOVA will also be performed to compare whether there are differences in R2*, ASL, HASTE, and BOLD signals between primary dysmenorrhea, endometriosis and leiomyoma participants.
Calculate response profiles of MRI signals associated with NSAID-resistance | through study completion, an average of 16 weeks
  Data will be processed similarly to Outcome #1. The investigators will use a repeated measures ANOVA and ANCOVA to examine changes in mean R2*, ASL, HASTE, or EPI-BOLD signal intensity (4 dependent variables) after naproxen and/or placebo administration in all women with primary dysmenorrhea-regardless of cluster identity or phenotype. The investigators will also use an ANCOVA to examine whether the 4 MRI metrics of uterine physiology are related to changes in pain, using the difference of VAS (Visual Analog Scale) after naproxen minus the VAS before naproxen as a covariate. The investigators will detect for ANCOVA assumptions (e.g., homogeneity of variance, normality) and utilize appropriate corrections (transformation, permutation analysis) when needed.
Calculate phenotype consistency | through study completion, an average of 16 weeks
  The investigators will also use a paired X2 (McNemar) test to establish reliability of the repeat scans and examine differences in cluster/phenotype categorization across visits. The combined use of principal component analysis, hierarchical testing, and validation by a repeatability test follows recommended guidelines

SECONDARY OUTCOMES:
Anatomical effects | through study completion, an average of 16 weeks
  Since participants with anatomical anomalies are provisionally excluded, the investigators will perform a sensitivity analysis by measuring the impact of provisional exclusion on linkage distance on clusters from Aim #1. Similarly, the impact of endometriosis and leiomyoma on cluster linkage distance will be calculated using recommended methods. Exploratory posthoc ANOVA/ANCOVAs will be performed within individual phenotypes/clusters identified in Aim #1 including endometriosis and leiomyoma to identify phenotypic-specific effects as a secondary analysis for Aim #2.
Covariate analysis | through study completion, an average of 16 weeks
  The investigators will calculate the correlation coefficient between NSAID resistance (defined as visual analog scale pain at 6 hours minus baseline pain) and age, parity, abuse (SPAQ score), anxiety (PROMIS Tscore), depression (PROMIS T-score), central pain sensitization (pain pressure thresholds). To accommodate differences in dimensionality we will use a combination of spearman, pearson, kendalls regression methods.
Calculate the relationship between Naproxen absorption and NSAID resistance. | through study completion, an average of 16 weeks
  The investigators will calculate the correlation coefficient between NSAID resistance (defined as visual analog scale pain at 6 hours minus baseline pain) and absorbed serum Naproxen (90 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Hellman, PhD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States